CLINICAL TRIAL: NCT00879008
Title: SYMPROVE III: Health Services Research Study for Treatment of the Moderate and Severe AECB
Brief Title: SYMPROVE III: Health Services Research Study for Treatment of the Moderate and Severe Acute Exacerbations of Chronic Bronchitis (AECB)
Acronym: SYMPROVE III
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 12629; AX0710DE (Other: Company Internal)
Record Dates: First submitted 2009-04-08; First posted 2009-04-09 (Estimated); Last update posted 2014-06-23 (Estimated); Status verified 2014-06

CONDITIONS: Chronic Bronchitis
Keywords: Disease Exacerbation; Acute Exacerbations of Chronic Bronchitis; AECB; Avelox; Bronchitis
MeSH Terms: conditions — Bronchitis, Chronic; Disease Progression; Bronchitis | interventions — Moxifloxacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Moxifloxacin (Avelox, BAY12-8039)

INTERVENTIONS:
Drug: Moxifloxacin (Avelox, BAY12-8039) — Patients from the normal praxis routine, treated with Moxifloxacin according to the local product information

SUMMARY:
In this study data of patients with moderate or severe acute exacerbations of chronic bronchitis (AECB) were collected. There were two different cohorts which were compared (Moxifloxacin and other antibiotics) concerning effectiveness and tolerance. It was a prospective study which was accomplished in 100 ambulatory practice offices.

DETAILED DESCRIPTION:
The study design was slightly changed to adapt the target population. Due to these changes the study was restarted on 8th December 2009.

ELIGIBILITY:
Inclusion Criteria:

* Acute exacerbation of chronic bronchitis from Anthonisen type I or II
* FEV1 of < 50 %
* Patient must be ensured in the statutory health insurance
* Further contraindications of the prescribed pharmaceutical products must be considered

Exclusion Criteria:

* Patients who change from one cohort to the other

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: It is a multicentre study in the ambulatory sector. Every primary care physician or pulmologist should inclose the first 5 patients with AECB from Anthonisen type I or II
Sampling Method: Non-Probability Sample
Enrollment: 345 (Actual)
Dates: Start 2009-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Effectiveness and tolerance of/to the different therapies | within the first 14 days
Possible hospitalisation rate | within the first 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Germany